CLINICAL TRIAL: NCT06270550
Title: Efficacy of Dynamic Movement Intervention on Children with Spastic Diplegia
Brief Title: Role of Dynamic Movement Intervention in Children with Spastic Diplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel Aziz Abdel Aziz Awara, Bachelor's degree in Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMI in Spastic Diplegia
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Spastic Diplegia
Keywords: Dynamic Movement Intervention
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic movement intervention based group. (Experimental)
  Interventions: Other: Dynamic Movement Intervention
- Selective physical therapy program based group. (Experimental)
  Interventions: Other: Dynamic Movement Intervention

INTERVENTIONS:
Other: Dynamic Movement Intervention — Dynamic movement intervention is a physical therapy approach for infants suffering abnormal developmental motor evolution caused by a known or unknown non-degenerative syndrome affecting the central nervous system

SUMMARY:
The study aims to investigate the effect of dynamic movement intervention approach on static and dynamic balance, quality of step length and cadence of walking pattern of children with spastic diplegic cerebral palsy.

ELIGIBILITY:
Inclusion criteria:

* Age ranged from 4-7 years.
* They can walk alone short distance and climb stairs holding on rail (Grade I & II according to GMFCS).
* They can understand and execute instructions.
* They will be medically stable.
* Degree of spasticity will be ranged from 1 to 1+ degree according to the Modified Ashworth Scale.

Exclusion criteria:

* Visual impairment (visual loss- cataract- myopia- hyperopia).
* Hearing impairment (deafness)
* Cognitive problem.
* Uncontrolled Convulsions.
* Orthopedic surgery for the affected lower limbs within one year.
* Botulinum toxin injection within the last 6 months or within the study period.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Dynamic movement intervention on balance and quality of walking of the study group compared to control group, measured using Humac Balance System. | Baseline
  Effect of Dynamic movement intervention on balance and quality of walking of the study group compared to control group with different intervention.
  As balance will be assessed using Humac Balance System.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No